CLINICAL TRIAL: NCT01090531
Title: A Multicenter, Prospective, Observational, Long-Term Follow-Up Study of Subjects With Chronic Hepatitis B and Low Viremia Who Do Not Receive Antiviral Therapy
Brief Title: Patients With Chronic Hepatitis B and Low Viremia Not Receiving Antiviral Therapy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Georg Dultz, MD, Johann Wolfgang Goethe University Hospital
Other Study IDs: JWGUHMED1-002
Record Dates: First submitted 2010-03-19; First posted 2010-03-22 (Estimated); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum
Oversight: Data Monitoring Committee: No

SUMMARY:
This observational long-term follow-up study will evaluate demographic, clinical, histological, biochemical, and virological parameters of patients with chronic hepatitis B and low viremia who do not require antiviral therapy according to current guidelines. Liver stiffness values as detected by FibroScan and ARFI will also be collected if available. All data will be collected at yearly intervals (minimum). Patients included in the study are followed for up to 10 years. The target sample size is <1000.

ELIGIBILITY:
Inclusion Criteria:

* adult patient, age 18-79
* chronic hepatitis B
* HBV-DNA < 100.000 IU/ml
* ALT ≤2 x ULN
* recent liver histology and/or FibroScan measurement
* willingness to sign informed consent

Exclusion Criteria:

* current or past antiviral therapy for hepatitis B
* chronic hepatitis B in immune tolerance phase (HBeAg positive, high viral load)
* co-infection with HIV, HCV
* malignant disease
* HCC or other liver tumor

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis B not receiving antiviral therapy
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2009-08; Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Indication for Antiviral Treatment | 10 years
Development of hepatocellular carcinoma (HCC) | 10 years
Progression of Liver Fibrosis | 10 years

SECONDARY OUTCOMES:
HBV-DNA | 10 years
Quantitative HBsAg | 10 years
Serum ALT | 10 years
Serum AFP | 10 years
FibroTest/ActiTest | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Sarrazin, MD, Principal Investigator — Medizinische Klinik 1, Klinikum der J. W. Goethe-Universität Frankfurt am Main, Germany
Locations (6):
- Germany (6):
  - Charité Berlin-Campus Virchow-Klinikum, Berlin
  - Klinikum der J. W. Goethe-Universität, Frankfurt
  - Institut für Interdisziplinäre Medizin, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Gastroenterologische Gemeinschaftspraxis Herne, Herne
  - Gastroenterologische Gemeinschaftspraxis Kiel, Kiel